CLINICAL TRIAL: NCT05821374
Title: Novel Treatment of Pyoderma Gangrenosum With Deucravacitinib
Brief Title: Deucravacitinib in PG
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Issues with funding and IND holder
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Brian.J.Simmons, Director of Dermatology Research, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02001753
Record Dates: First submitted 2023-03-20; First posted 2023-04-20 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — deucravacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Deucravacitinib (Experimental): Participants to receive Deucravacitinib 6 mg tablets orally twice daily for 12 weeks.
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — 6 mg tablet
  Other Names: SOTYKTU

SUMMARY:
The main goal of this study is to see if the study drug called "Deucravacitinib" is safe and effective in treating people with pyoderma gangrenosum (PG).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18-70 years old
* Diagnosed with pyoderma gangrenosum requiring one major and at least 4 minor criteria
* Women must not be pregnant, lactating, or planning pregnancy during the study period
* Women of child-bearing potential must be on birth control for the duration of the treatment period.
* Subjects must agree to the use of at least one of the following contraception methods for the entire duration of the study until at least 30 days after taking their last dose of study drug:
* Women: Hormonal contraception (oral, injections, patch, implant, or vaginal-ring); Spiral (with or without hormones); any sterilization methods; a partner who has had a vasectomy; or sexual abstinence.
* Other acceptable methods of contraception are male or female condoms (with or without spermicide) or a cap, diaphragm, or sponge with spermicide.
* Willing to discontinue topical and/or systemic therapies, with the exception of oral rescue therapy with steroids.
* The wash period for systemic therapies will largely depend on the specific treatment but, in general, will be at least 6 months for biologics and 3 months for other immune- suppressants such as cyclosporine, mycophenolate mofetil, methotrexate, etc. No wash out period is required for topicals.
* Capable and willing to sign Institutional Review Board/IEC-approved written informed consent form in accordance with regulatory and institutional guidelines before the performance of any protocol-related procedures.

Exclusion Criteria:

* Patient under 18 years of age.
* Patients with a history of inflammatory bowel disease.
* Patients on systemic immunosuppressive/immune modulating therapy including: oral steroids, cyclosporine, mycophenolate mofetil, methotrexate, Azathioprine or TNFα inhibitor at time of starting deucravacitinib.
* Patients currently enrolled in another investigational study.
* Patients with a history or evidence of active infection and/or febrile illness within 7 days; or serious infection requiring antibiotic treatment within 30 days
* Hepatitis C virus (HCV): subjects known to be positive for anti-HCV antibody or for HCV RNA detectable by polymerase chain reaction (PCR)
* Hepatitis B virus (HBV): subjects known to be positive for hepatitis B surface antigen or for HBV DNA detectable by PCR
* Human Immunodeficiency Virus (HIV) infection: subjects known to be HIV positive
* History of active or inadequately treated latent tuberculosis (TB)
* Known or suspected systemic or skin autoimmune disorder other than pyoderma gangrenosum
* Any unstable major illness or evidence of unstable condition of major organ systems including psychiatric
* Cancer or history of lymphoproliferative disease within last 5 years; exception is cutaneous basal cell carcinoma or squamous cell carcinoma that has been treated.
* Major surgery within the last 4 weeks
* Live vaccines within the last 60 days
* Leukopenia (absolute WBC count < 3000/mm3); Lymphopenia (ALC < 500/mm3); Neutropenia (ANC < 1000/mm3)
* Thrombocytopenia (platelet count < 100,000/mm3; Anemia (hemoglobin < 9.0g/dL)
* ALT/AST > 3 X ULN and/or Total, unconjugated, and/or conjugated bilirubin > 2 X ULN within 28 days of dosing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Change in Physician's Global Assessment (PGA) | Baseline; Days 8, 15, 29, 57, and 85; Follow up Day 115
  PGA will be used for overall assessment of efficacy.
Change from baseline in ulcer size measured by calculating the area of the ulcers in centimeters squared using a digital application. | Baseline; Days 8, 15, 29, 57, and 85; Follow up Day 115
  imitoAG application for mobile devices will be used to calculate the dimensions of the ulcers in centimeters to determine if the size of the ulcers is changed by the treatment.

SECONDARY OUTCOMES:
The percentage of patients needing rescue therapy from baseline to Day 115 | Baseline through Day 115
  Determining the number of participants that required rescue therapy while on study.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Simmons, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No